CLINICAL TRIAL: NCT03701997
Title: All-comers Registry Monitoring the Safety and Effectiveness of the Berlin Heart EXCOR® Pediatric VAD as a Bridge to Cardiac Transplantation.
Brief Title: Registry to Monitor Berlin Heart EXCOR® Pediatric VAD as a Bridge to Cardiac Transplantation.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Berlin Heart, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EXCOR PMA Post Approval
Record Dates: First submitted 2018-10-09; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Ventricular Dysfunction; Ventricular Dysfunction, Left; Ventricular Dysfunction, Right
MeSH Terms: conditions — Ventricular Dysfunction; Ventricular Dysfunction, Left; Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes

GROUPS / COHORTS (1):
- EXCOR Pediatric: Pediatric (age 0 - 21) patients who are transplant eligible in need of mechanical circulatory support and are supported with the EXCOR® Pediatric
  Interventions: Device: EXCOR Pediatric

INTERVENTIONS:
Device: EXCOR Pediatric — Mechanical circulatory support using ventricular assist device
  Other Names: EXCOR Pediatric VAD; EXCOR Pediatric Ventricular Assist Device; Berlin Heart EXCOR Pediatric; EXCOR

SUMMARY:
The purpose of this post market surveillance is to continue monitoring the safety and effectiveness of the Berlin Heart EXCOR® Pediatric. This surveillance includes an "all-comers" prospective cohort of pediatric (<22 years of age) patients implanted according to the IFU with the EXCOR® Pediatric.

DETAILED DESCRIPTION:
The Advanced Cardiac Therapies Improving Outcomes Network (Action) database will be used for the surveillance. The network was developed to determine best practice and improve quality in the pediatric mechanical circulatory support field. The registry Protocol and Manual of Operations will be followed by participating pediatric transplant hospitals. Quality assurance of the data will be monitored by the registry's data coordinating center.

ELIGIBILITY:
Inclusion Criteria:

* Transplant eligible
* Implanted with EXCOR Pediatric per IFU

Exclusion Criteria:

* Having any contradictions for user per IFU

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric (0-21 years) who are transplant eligible in need of mechanical circulatory support and are supported with the EXCOR® Pediatric
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Stroke rate | Until discontinuation of device support or 180 days
  The primary endpoint is to demonstrate that the rate of stroke (ischemic or hemorrhagic) will be no worse than the pre-specified performance goal. The rate will be calculated as the proportion of subjects experiencing a stroke while on EXCOR® Pediatric support within the first 180 days post-implant. The upper bound of the 95% confidence interval for the observed stroke rate will be compared to the pre-specified performance goal of 30%.

SECONDARY OUTCOMES:
Adverse Events | Until discontinuation of device support or 180 days
  Adverse Event rates per patient-month
Device effectiveness | Until discontinuation of device support or 180 days
  Proportion of subjects experiencing a successful (transplant, wean for recovery) outcome

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kroslowitz, BS, Study Director — Berlin Heart, Inc
Locations (1):
- Sites per Action network, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No